CLINICAL TRIAL: NCT00129961
Title: A Randomized, Open-Label Study to Compare the Rate of New Non-Melanoma Skin Cancer in Maintenance Renal Allograft Recipients Converted to a Sirolimus-based Regimen Versus Continuation of a Calcineurin Inhibitor-based Regimen
Brief Title: Study Evaluating the Effect of Sirolimus on Non-Melanoma Skin Cancer in Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0468H1-407
Record Dates: First submitted 2005-08-01; First posted 2005-08-12 (Estimated); Results first posted 2012-03-23 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Skin Neoplasms; Kidney Transplantation
Keywords: Kidney; Transplant; Skin Cancer
MeSH Terms: conditions — Skin Neoplasms | interventions — Sirolimus; Cyclosporine; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Conversion to a sirolimus-based regimen
  Interventions: Drug: sirolimus
- 2 (Active Comparator): Continuation of a CNI-based regimen
  Interventions: Drug: cyclosporine or tacrolimus

INTERVENTIONS:
Drug: sirolimus
  Arms: 1
Drug: cyclosporine or tacrolimus
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effect of sirolimus on the prevention of new non-melanoma skin cancer (NMSC) in kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant at least 1 year prior
* Subjects with a functioning renal allograft with calculated glomerular filtration rate (GFR) ≥40mL/min (Nankivell method) and proteinuria ≤500mg/day.
* Stable on cyclosporine or tacrolimus-based multi-drug immunosuppressive regimen
* History of NMSC within last 3 years

Exclusion Criteria:

* History of other cancer within last 3 years
* NMSC with metastatic disease or more than 20 NMSC lesions in last 12 months
* Multiple organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2005-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Canada, clintrialparticipation@wyeth.com; Trial Manager, Principal Investigator — For Australia, medinfo@wyeth.com; Trial Manager, Principal Investigator — For New Zealand, medinfo@wyeth.com
Locations (23):
- United States (12):
  - San Diego, California
  - San Francisco, California
  - Gainesville, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee
  - Madison, Wisconsin
- Australia (9):
  - Camperdown, New South Wales
  - Wooloongabba, Queensland
  - Woodville, South Australia
  - Adelaide
  - Clayton
  - Herston
  - Parkville
  - Randwick
  - Westmead
- Vancouver, British Columbia, Canada
- Grafton, Auckland, New Zealand

REFERENCES:
- [Derived] Campbell SB, Walker R, Tai SS, Jiang Q, Russ GR. Randomized controlled trial of sirolimus for renal transplant recipients at high risk for nonmelanoma skin cancer. Am J Transplant. 2012 May;12(5):1146-56. doi: 10.1111/j.1600-6143.2012.04004.x. Epub 2012 Mar 15. PMID 22420843

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in Australia, New Zealand and North America from August 2005 (first subject randomized September 2005) through October 2007.
Pre-assignment Details: Screening and baseline evaluations were performed within 4 weeks prior to randomization. Randomization assignments by site were stratified by the number of new NMSC lesions in the 12 months prior to enrollment (0-5 lesions vs 6-20 lesions).
Groups:
- Sirolimus (SRL) Based Regimen: All subjects discontinued Calcineurin inhibitors (CNI) after the morning dose on day 1. SRL was initiated with a loading dose of 6-12mg on day 1, followed by 2-4mg daily and was adjusted to maintain a whole blood trough concentration of 5-15ng/mL (high performance liquid chromatography [HPLC]). Once the SRL trough concentration was ≥ 5ng/mL, subjects receiving mycophenolate mofetil (MMF), mycophenolate sodium (MPS), or azathioprine (AZA) at randomization had doses reduced to ≤1.5 g/day, ≤1080 mg/day or ≤75 mg/day respectively. If warranted subjects could be switched between MMF, MPS, or AZA or their doses decreased, temporarily withheld, or discontinued. Subjects receiving corticosteroids (CS) at time of randomization or if MMF, MPS, or AZA was discontinued, had to receive CS ≥2.5mg/day of prednisone. Subjects not receiving MMF, MPS, or AZA at time of randomization remained on a minimum of double therapy (SRL and CS). Addition of MMF, MPS, or AZA was permitted.
- Calcineurin Inhibitor (CNI) Based Regimen: Baseline CNI therapy was continued after randomization and doses could be adjusted throughout the study as indicated, but therapy could not be withdrawn. Cyclosporine could be switched to tacrolimus, and vice versa. If warranted subjects could be switched between MMF, MPS, or AZA or their doses could be decreased, temporarily withheld, or discontinued. Subjects undergoing discontinuation of MMF, MPS, or AZA had to receive CS ≥2.5 mg/day of prednisone or the equivalent thereof. If subjects were not receiving MMF, MPS, or AZA at the time of randomization, the addition of MMF, MPS, or AZA was permitted if clinically indicated. If subjects were receiving CS at the time of randomization, CS was maintained at ≥2.5 mg/day of prednisone or the equivalent thereof. CS withdrawal was prohibited. If subjects were not receiving CS at the time of randomization, treatment could be initiated during the conduct of the study if clinically indicated.
Period: Overall Study
Arm/Group | Sirolimus (SRL) Based Regimen | Calcineurin Inhibitor (CNI) Based Regimen
Started | 39 | 47
Completed | 20 | 24
Not Completed | 19 | 23
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 1
Not completed — Withdrawal by Sponsor | 14 | 20
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Missing Record | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sirolimus (SRL) Based Regimen | Calcineurin Inhibitor (CNI) Based Regimen | Total
Number analyzed (Participants) | 39 | 47 | 86
Age Continuous [Mean (Full Range); unit: years] | 59.08 [36 to 76] | 58.98 [37 to 78] | 59.02 [36 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 31 | 34 | 65
Stratification Group [Number; unit: subjects]
  0-5 Lesions in 12 months prior | 33 | 39 | 72
  6-20 Lesions in 12 months prior | 6 | 8 | 14
Time from Current Transplantation to Randomization [Mean (Standard Deviation); unit: Months] | 114.98 (57.63) | 109.57 (55.08) | 112.02 (55.98)

OUTCOME MEASURES:

1. Primary Outcome: New Biopsy-Confirmed Nonmelanoma Skin Cancer (NMSC) Lesions Per Subject Per Year
Description: The number of new biopsy-confirmed NMSC lesions per subject per year was calculated by summarizing the total number of new BCC and SCC lesions reported over the observation period and standardizing it to an annual rate by multiplying by 365 and dividing by days on study.
Time Frame: up to 24 months
Population: Intention to Treat: All randomly assigned subjects with at least 1 dose of study medication, includes data of subjects on therapy, those off therapy, and those who completed follow-up.
Measure: Number; unit: Standardized Yearly Rate of NMSC
Arm/Group | Sirolimus (SRL) Based Regimen | Calcineurin Inhibitor (CNI) Based Regimen
Number analyzed (Participants) | 39 | 47
Standardized Yearly Rate of NMSC | 1.31 (0.52) | 2.48 (0.69)
Statistical Analysis 1: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; Test type: Superiority or Other; p = 0.022, Poisson regression — Poisson regression was used to model NMSC counts using the years in study as an offset. The generalized estimated equations (GEE) approach was used to estimate parameters and compare treatment differences; Adjusted by baseline strata; Poisson model = strata + treatment

2. Secondary Outcome: Time to First Biopsy Confirmed New NMSC Lesion.
Description: The time to first biopsy confirmed new NMSC lesion starts at 1 day post randomization to biopsy and/or treatment of newly confirmed NMSC lesion.
Time Frame: up to 24 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: number of days
Arm/Group | Sirolimus (SRL) Based Regimen | Calcineurin Inhibitor (CNI) Based Regimen
Number analyzed (Participants) | 39 | 47
number of days | 380 (42.42) [227 to NA] — Upper limit for 95% CI is not available because the curve representing the upper CI limit for the survivor function lies above 0.5 (or where the horizontal line at 50% does not intersect a CI), the upper CI limit for the median cannot be estimated. | 163 (42.32) [96 to 253]
Statistical Analysis 1: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; Test type: Superiority or Other; p = 0.047, Regression, Cox; Stratified by baseline lesions

3. Secondary Outcome: Number of Lesion Free Subjects
Description: The overall number of subjects who were lesion free were compared between treatment groups with the Cochran Mantel Haenszel test stratified by baseline NMSC stratum. Within each stratum, the Fisher exact test was used to compare the proportions of lesion free subjects between treatment groups.
Time Frame: up to 24 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sirolimus (SRL) Based Regimen | Calcineurin Inhibitor (CNI) Based Regimen
Number analyzed (Participants) | 39 | 47
participants | 17 | 9
Statistical Analysis 1: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; Test type: Superiority or Other; p = 0.015, Cochran-Mantel-Haenszel; Stratified by baseline lesion strata

4. Secondary Outcome: Percentage of Patients With New Biopsy-confirmed NMSC: Squamous Cell Carcinoma (SCC) and Basal Cell Carcinoma (BCC)
Time Frame: up to 24 months
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Sirolimus (SRL) Based Regimen | Calcineurin Inhibitor (CNI) Based Regimen
Number analyzed (Participants) | 39 | 47
Percentage of Participants
  SCC | 67 | 69
  BCC | 33 | 31
Statistical Analysis 1: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; Test type: Superiority or Other; p = 0.799, Chi-squared

5. Secondary Outcome: Grade Distribution of NMSC Lesions
Description: Number of subjects with at least 1 biopsy-confirmed new squamous cell carcinoma (SCC) or basal cell carcinoma (BCC).
Time Frame: up to 24 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sirolimus (SRL) Based Regimen | Calcineurin Inhibitor (CNI) Based Regimen
Number analyzed (Participants) | 39 | 47
participants
  SCC Well differentiated | 5 | 17
  SCC Moderately differentiated | 9 | 14
  SCC Poorly differentiated | 1 | 1
  SCC Invasive | 10 | 24
  SCC In Situ | 12 | 27
  SCC Invasive with Perineural Invasion | 2 | 1
  SCC Invasive without Perineural Invasion | 8 | 24
  BCC Superficial | 7 | 16
  BCC Nodular | 11 | 15
  BCC Infiltrative | 2 | 6
Statistical Analysis 1: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; SCC Well differentiated; Test type: Superiority or Other; p = 0.014, Cochran-Mantel-Haenszel; Stratified by baseline lesion strata
Statistical Analysis 2: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; SCC Moderately differentiated; Test type: Superiority or Other; p = 0.491, Cochran-Mantel-Haenszel; Stratified by baseline lesion strata
Statistical Analysis 3: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; SCC Poorly differentiated; Test type: Superiority or Other; p = 0.905, Cochran-Mantel-Haenszel; Stratified by baseline lesion strata
Statistical Analysis 4: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; SCC Invasive; Test type: Superiority or Other; p = 0.018, Cochran-Mantel-Haenszel; Stratified by baseline lesion strata
Statistical Analysis 5: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; SCC In Situ; Test type: Superiority or Other; p = 0.012, Cochran-Mantel-Haenszel; Stratified by baseline lesion strata
Statistical Analysis 6: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; SCC Invasive with Perineural Invasion; Test type: Superiority or Other; p = 0.463, Cochran-Mantel-Haenszel; Stratified by baseline lesion strata
Statistical Analysis 7: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; SCC Invasive without Perineural Invasion; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel; Stratified by baseline lesion strata
Statistical Analysis 8: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; BCC Superficial; Test type: Superiority or Other; p = 0.094, Cochran-Mantel-Haenszel; Stratified by baseline lesion strata
Statistical Analysis 9: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; BCC Nodular; Test type: Superiority or Other; p = 0.720, Cochran-Mantel-Haenszel; Stratified by baseline lesion strata
Statistical Analysis 10: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; BCC Infiltrative; Test type: Superiority or Other; p = 0.227, Cochran-Mantel-Haenszel; Stratified by baseline lesion strata

6. Secondary Outcome: Number of Recurrent NMSC Lesions Per Subject-year
Description: Recurrent NMSC lesions is defined as recurring at the site of a previously treated lesion.
Time Frame: up to 24 months
Population: as for outcome 1
Measure: Number; unit: lesions per participant year
Arm/Group | Sirolimus (SRL) Based Regimen | Calcineurin Inhibitor (CNI) Based Regimen
Number analyzed (Participants) | 39 | 47
lesions per participant year | 0.107 (0.09) | 0.134 (0.10)
Statistical Analysis 1: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; Test type: Superiority or Other; p = 0.748, Poisson regression

7. Secondary Outcome: Subjects Reporting Incidence of Metastatic Disease Related to NMSC.
Description: The number of subjects with metastatic disease related to NMSC.
Time Frame: up to 24 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sirolimus (SRL) Based Regimen | Calcineurin Inhibitor (CNI) Based Regimen
Number analyzed (Participants) | 39 | 47
participants | 1 | 3
Statistical Analysis 1: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; Test type: Superiority or Other; p = 0.425, Cochran-Mantel-Haenszel; Stratified by baseline lesion strata

8. Secondary Outcome: Death Due to NMSC
Time Frame: up to 24 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sirolimus (SRL) Based Regimen | Calcineurin Inhibitor (CNI) Based Regimen
Number analyzed (Participants) | 39 | 47
participants | 0 | 0

9. Secondary Outcome: Number of Subjects Who Discontinue Assigned Therapy
Time Frame: up to 24 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sirolimus (SRL) Based Regimen | Calcineurin Inhibitor (CNI) Based Regimen
Number analyzed (Participants) | 39 | 47
participants | 31 | 23

10. Secondary Outcome: Nankivell-Calculated Glomerular Filtration Rate (GFR)
Description: GFR is an index of kidney function. GFR describes the flow rate of filtered fluid through the kidney. GFR can be measured directly or estimated using established formulas. For this study, GFR was calculated using Nankivell. A normal GFR is > 90 mL/min, although children and older people usually have a lower GFR. Lower values indicate poor kidney function. A GFR <15 is consistent with kidney failure.
Time Frame: At 24 months (week 104)
Population: Intention to Treat: All randomly assigned subjects with at least 1 dose of study medication, includes data of subjects on therapy, those off therapy, and those who completed follow-up. For the intention to treat analysis, a GFR of 0 was imputed for graft loss or death, and last observation carried forward (LOCF) for missing values.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Sirolimus (SRL) Based Regimen | Calcineurin Inhibitor (CNI) Based Regimen
Number analyzed (Participants) | 39 | 47
units on scale | 72.49 (24.41) | 68.42 (19.91)
Statistical Analysis 1: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; Test type: Superiority or Other; p = 0.604, ANCOVA

11. Secondary Outcome: Serum Creatinine Level
Description: Serum creatinine is an indicator of kidney function. Creatinine is a substance formed from the metabolism of creatinine, commonly found in blood, urine, and muscle tissue. It is removed from the blood by the kidneys and excreted in urine. An increased level of creatinine in the blood indicates decreased kidney function. Normal adult blood levels of creatinine are 0.5 to 1.1 mg/dL for females and 0.6 to 1.2 mg/dL for males, however the normal values are age-dependent as elderly patients typically have smaller muscle mass.
Time Frame: At 24 months (Week 104)
Population: Intention to Treat: All randomly assigned subjects with at least 1 dose of study medication, includes data of subjects on therapy, those off therapy, and those who completed follow-up. All available data, no imputations.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Sirolimus (SRL) Based Regimen | Calcineurin Inhibitor (CNI) Based Regimen
Number analyzed (Participants) | 17 | 22
μmol/L | 139.35 (41.63) | 135.23 (37.84)
Statistical Analysis 1: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; Test type: Superiority or Other; p = 0.672, ANCOVA

12. Secondary Outcome: Number of Participants That Died
Time Frame: up to 24 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sirolimus (SRL) Based Regimen | Calcineurin Inhibitor (CNI) Based Regimen
Number analyzed (Participants) | 39 | 47
participants | 1 | 1
Statistical Analysis 1: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; Test type: Superiority or Other; p = 0.999, Fisher Exact

13. Secondary Outcome: Graft Survival Measured by Graft Loss
Description: Graft loss was defined as physical loss (nephrectomy), functional loss (necessitating maintenance dialysis for >8 consecutive weeks), retransplant, or death.
Time Frame: up to 24 months
Population: as for outcome 1
Measure: Number; unit: graft loss
Arm/Group | Sirolimus (SRL) Based Regimen | Calcineurin Inhibitor (CNI) Based Regimen
Number analyzed (Participants) | 39 | 47
graft loss | 2 | 1
Statistical Analysis 1: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; Test type: Superiority or Other; p = 0.588, Fisher Exact

14. Secondary Outcome: Number of Subjects With Biopsy-Confirmed Acute Rejection
Time Frame: up to 24 months
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Sirolimus (SRL) Based Regimen | Calcineurin Inhibitor (CNI) Based Regimen
Number analyzed (Participants) | 39 | 47
subjects | 0 | 1
Statistical Analysis 1: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; Test type: Superiority or Other; p = 0.999, Fisher Exact

15. Secondary Outcome: Spot Urine Protein:Creatinine Ratio
Description: Subjects' urine protein:creatinine ratios were summarized by each scheduled visit, and the nonparametric Wilcoxon rank sum test was used to compare the difference between groups.
Time Frame: At 24 months (Week 104)
Population: Intention to Treat: All randomly assigned subjects with at least 1 dose of study medication, includes data of subjects on therapy, those off therapy, and those who completed follow-up. Available data, no imputations.
Measure: Median (Full Range); unit: ratio (mg/mg)
Arm/Group | Sirolimus (SRL) Based Regimen | Calcineurin Inhibitor (CNI) Based Regimen
Number analyzed (Participants) | 13 | 22
ratio (mg/mg) | 0.14 (0.28) [0.09 to 1.07] | 0.12 (0.08) [0.04 to 0.34]
Statistical Analysis 1: Comparison: Sirolimus (SRL) Based Regimen vs Calcineurin Inhibitor (CNI) Based Regimen; Test type: Superiority or Other; p = 0.030, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Sirolimus (SRL) Based Regimen | Calcineurin Inhibitor (CNI) Based Regimen
Serious Adverse Events (participants affected / at risk) | 15/39 | 21/47
Other Adverse Events (participants affected / at risk) | 38/39 | 40/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus (SRL) Based Regimen (N=39) | Calcineurin Inhibitor (CNI) Based Regimen (N=47)
Allergic reaction (General disorders) | 1 | 0
Cellulitis (General disorders) | 1 | 1
Neoplasm (General disorders) | 0 | 1
Sepsis (General disorders) | 0 | 3
Transplant rejection (General disorders) | 1 | 1
Aneurysm (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Arterial anomaly (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Deep vein thrombosis (Cardiac disorders) | 0 | 1
Heart failure (Cardiac disorders) | 1 | 0
Hypertension (Cardiac disorders) | 1 | 0
Left heart failure (Cardiac disorders) | 1 | 0
Myocardial infarct (Cardiac disorders) | 1 | 0
Thrombosis (Cardiac disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 3
Nausea and vomiting (Gastrointestinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 1
Lymphoma (Blood and lymphatic system disorders) | 1 | 0
Creatinine increased (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Confusion (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Subdural hematoma (Metabolism and nutrition disorders) | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Metabolism and nutrition disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin carcinoma (Skin and subcutaneous tissue disorders) | 1 | 2
Skin melanoma (Skin and subcutaneous tissue disorders) | 0 | 2
Acute kidney failure (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Kidney failure (Renal and urinary disorders) | 1 | 0
Prostatic carcinoma (Renal and urinary disorders) | 2 | 1
Pyelonephritis (Renal and urinary disorders) | 0 | 1
Urinary tract infection (Renal and urinary disorders) | 1 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus (SRL) Based Regimen (N=39) | Calcineurin Inhibitor (CNI) Based Regimen (N=47)
Abdominal Pain (General disorders) | 1 | 5
Accidental Injury (General disorders) | 4 | 5
Adenoma (General disorders) | 0 | 1
Allergic reaction (General disorders) | 3 | 0
Asthenia (General disorders) | 2 | 0
Back pain (General disorders) | 0 | 2
Chest pain (General disorders) | 4 | 2
Cyst (General disorders) | 1 | 2
Drug level decreased (General disorders) | 0 | 1
Drug level increased (General disorders) | 2 | 0
Face edema (General disorders) | 1 | 0
Fever (General disorders) | 1 | 1
Flu syndrome (General disorders) | 1 | 0
Headache (General disorders) | 5 | 1
Hernia (General disorders) | 1 | 0
Hormone level altered (General disorders) | 0 | 1
Infection (General disorders) | 0 | 1
Lab test abnormal (General disorders) | 2 | 1
Malaise (General disorders) | 1 | 0
Neck pain (General disorders) | 0 | 1
Neoplasm (General disorders) | 0 | 2
Pain (General disorders) | 6 | 5
Pelvic pain (General disorders) | 1 | 3
Tolerance decreased (General disorders) | 2 | 0
Transplant rejection (General disorders) | 0 | 1
Aneurysm (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Arterial anomaly (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiomegaly (Cardiac disorders) | 0 | 1
Cardiovascular physical finding (Cardiac disorders) | 2 | 1
Cyanosis (Cardiac disorders) | 0 | 1
Deep vein thrombosis (Cardiac disorders) | 0 | 1
Heart failure (Cardiac disorders) | 1 | 0
Hemorrhage (Cardiac disorders) | 0 | 1
Hypertension (Cardiac disorders) | 6 | 4
Hypotension (Cardiac disorders) | 0 | 3
Left heart failure (Cardiac disorders) | 1 | 0
Myocardial infarct (Cardiac disorders) | 1 | 0
Peripheral vascular disorder (Cardiac disorders) | 0 | 1
Retinal artery occlusion (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 1
Thrombophlebitis superficial (Cardiac disorders) | 0 | 1
Thrombosis (Cardiac disorders) | 0 | 1
Anorexia (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhea (Gastrointestinal disorders) | 16 | 6
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Fecal incontinence (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2
Gastroenteritis (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 3
Liver fatty deposit (Gastrointestinal disorders) | 0 | 1
Liver function tests abnormal (Gastrointestinal disorders) | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 13 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Rectal disorder (Gastrointestinal disorders) | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 2 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 0
Tongue discoloration (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3
Thyroid disorder (Endocrine disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 4 | 2
Antinuclear antibody present (Blood and lymphatic system disorders) | 1 | 0
Ecchymosis (Blood and lymphatic system disorders) | 2 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Avitaminosis (Metabolism and nutrition disorders) | 0 | 1
Creatinine increased (Metabolism and nutrition disorders) | 2 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Edema (Metabolism and nutrition disorders) | 1 | 0
Glucose tolerance decreased (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 5 | 3
Hypercholesteremia (Metabolism and nutrition disorders) | 3 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0
Hyperlipemia (Metabolism and nutrition disorders) | 5 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Lactic dehydrogenase increased (Metabolism and nutrition disorders) | 0 | 1
Peripheral edema (Metabolism and nutrition disorders) | 16 | 3
Sgpt increased (Metabolism and nutrition disorders) | 0 | 1
Thirst (Metabolism and nutrition disorders) | 1 | 0
Weight loss (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Depression (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 3
Dizziness postural (Nervous system disorders) | 0 | 2
Emotional lability (Nervous system disorders) | 1 | 0
Hypesthesia (Nervous system disorders) | 0 | 1
Insomnia (Nervous system disorders) | 1 | 0
Nervousness (Nervous system disorders) | 1 | 0
Neuropathy (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 2 | 0
Sleep disorder (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 2 | 1
Subdural hematoma (Nervous system disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough increased (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration nos (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 7 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 3 | 0
Folliculitis (Skin and subcutaneous tissue disorders) | 3 | 1
Fungal dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Herpes simplex (Skin and subcutaneous tissue disorders) | 1 | 1
Herpes zoster (Skin and subcutaneous tissue disorders) | 1 | 1
Maculopapular rash (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritic rash (Skin and subcutaneous tissue disorders) | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Pustular rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 13 | 1
Seborrheic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin carcinoma (Skin and subcutaneous tissue disorders) | 1 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 3
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 2 | 4
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Abnormal vision (Eye disorders) | 1 | 0
Cataract specified (Eye disorders) | 2 | 2
Conjunctivitis (Eye disorders) | 1 | 0
Dry eyes (Eye disorders) | 1 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Eye disorder (Eye disorders) | 1 | 1
Eye hemorrhage (Eye disorders) | 2 | 0
Otitis media (Ear and labyrinth disorders) | 0 | 1
Retinal disorder (Eye disorders) | 1 | 0
Retinal edema (Eye disorders) | 1 | 0
Taste perversion (Gastrointestinal disorders) | 2 | 0
Acute kidney failure (Renal and urinary disorders) | 1 | 1
Albuminuria (Renal and urinary disorders) | 7 | 0
Breast disorder (Reproductive system and breast disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 3
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Hydroureter (Renal and urinary disorders) | 1 | 0
Kidney function abnormal (Renal and urinary disorders) | 0 | 1
Prostatic specific antigen increase (Renal and urinary disorders) | 0 | 1
Testis disorder (Renal and urinary disorders) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Urogenital disorder (Renal and urinary disorders) | 1 | 0
Allergic reaction other than drug (General disorders) | 0 | 1
Device malfunction (General disorders) | 1 | 0
Local reaction to procedure (General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
A blinded review of data in May 2007 determined there was minimal added power in follow-up through 2 years vs. 1 year. The study was then amended to require at least 1 year of follow-up instead of 2 years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.